CLINICAL TRIAL: NCT07172022
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, Multicenter Study Evaluating Efficacy, Safety, and Pharmacokinetics of Crovalimab in Patients With Antiphospholipid Syndrome (APS)
Brief Title: A Study to Evaluate Crovalimab in People With Antiphospholipid Syndrome (APS)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO46107; 2025-522980-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-11; First posted 2025-09-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crovalimab + VKA (Experimental): Participants will receive 3 loading doses of crovalimab, 680 milligrams (mg) or 1020 mg, as a subcutaneous (SC) injection based on their body weight (BW) at Weeks 1, 2 and 3 followed by maintenance doses, every 4 weeks (Q4W) from Week 5 until arterial thrombosis, venous thromboembolism or cardiovascular death. Participants will also receive VKA with a target internal normalized ratio (INR) based on investigator's discretion and local guidance.
  Interventions: Drug: Crovalimab; Drug: VKA
- Placebo + VKA (Placebo Comparator): Participants will receive 3 doses of placebo as a SC injection with equal volume dosing as the weight-based crovalimab at Weeks 1, 2, and 3, followed by Q4W doses, as a SC injection, from Week 5 until arterial thrombosis, venous thromboembolism, or cardiovascular death. Participants will also receive VKA with a target INR based on the investigator's discretion and local guidance.
  Interventions: Drug: Placebo; Drug: VKA

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 680 mg (for participants with BW ≥ 40 kilograms [kg] to < 100 kg) or 1020 mg (for participants with BW ≥ 100 kg), as a SC injection, at Weeks 1, 2, and 3 and Q4W from Week 5 onwards.
  Other Names: RO7112689; SKY59; PIASKY
  Arms: Crovalimab + VKA
Drug: Placebo — Placebo matching crovalimab will be administered as per the schedule specified in the respective arm.
  Arms: Placebo + VKA
Drug: VKA — Dose administration of VKA will be in accordance with the local prescribing information for the respective product. The VKA regimen will be titrated to a therapeutic target INR based on investigator discretion and local standard of care (SOC).

SUMMARY:
The main purpose of this study is to evaluate the efficacy of crovalimab compared with placebo as an add-on therapy to vitamin K antagonist (VKA) in participants with APS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤70 years, and body weight ≥40 kilograms (kg), at the time of signing Informed Consent Form
* Vaccination against N. meningitidis, H. influenzae type B, and S. pneumoniae
* Participants classified with APS who have experienced at least two prior arterial and/or venous thrombotic events, based on the 2023 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) criteria, positive for at least two of the following: lupus anticoagulant (LAC) test, anticardiolipin antibodies (aCL), anti-β2-glycoprotein 1 antibodies (aβ2GP1)
* Participants receiving corticosteroids, antimalarial treatment, non-biologic disease-modifying rheumatic drugs, statins, and low dose aspirin must be on a stable dose prior to the first dose of study treatment
* Willingness and ability to comply with a VKA regimen titrated to a therapeutic target internal normalized ratio (INR)
* Agreement to adhere to the contraception requirements

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant during the study or within the time frame in which contraception is required
* Treatment with investigational therapy, complement inhibitor, and/or other immune-suppressive biologic therapy within 5 half-lives of that agent prior to screening visit, or plans to participate in another investigational trial
* Presence of another systemic autoimmune disease that is unstable and requires additional treatment, and constitutes the principal illness and may impact evaluation of the concurrent APS
* Inadequate renal and hepatic function
* Uncontrolled hyperlipidemia and/or hypertension, known diabetes mellitus, and/or serious infection requiring hospitalization or antibiotics prior to Week 1 Day 1
* History or condition associated with increased bleeding risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2030-03-11 (Estimated); Study Completion 2030-12-02 (Estimated)

PRIMARY OUTCOMES:
Time From Randomization to First Occurrence of Objectively Confirmed Arterial Thrombosis, Venous Thromboembolism or Cardiovascular Death | Up to approximately 4.5 years

SECONDARY OUTCOMES:
Time From Randomization to the First Occurrence of Objectively Confirmed Venous Thromboembolism | Up to approximately 4.5 years
Time From Randomization to the First Occurrence of Objectively Confirmed Arterial Thrombosis | Up to approximately 4.5 years
Percentage of Participants With Adverse Events (AEs) With Severity Determined According to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) | Up to approximately 4.5 years
Percentage of Participants With Injection Site Reactions and Hypersensitivity | Up to approximately 4.5 years
Percentage of Participants With Infections and Severity of Infection | Up to approximately 4.5 years
Percentage of Participants With AEs Leading to Study Drug Discontinuation | Up to approximately 4.5 years
Serum Concentrations of Crovalimab Over Time | Up to approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing